CLINICAL TRIAL: NCT00749203
Title: Ketamine as a Rapid Treatment for Post-traumatic Stress Disorder
Brief Title: Ketamine as a Rapid Treatment for Post-traumatic Stress Disorder (PTSD)
Acronym: KetPTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dennis Charney (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Dennis Charney, Dean, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 07-1199; PT074949; IF1554104; A-15236 (Other: USAMRMC ORP HRPO)
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Stress Disorders, Post-Traumatic; PTSD; Depression; Anxiety Disorder
Keywords: Stress Disorders, Post-Traumatic; PTSD; anxiety disorder; ketamine; depression; depressed mood
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Consciousness Disorders | interventions — Midazolam; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Single dose 0.5 mg/kg IV (in the vein) infused over 40 minutes
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): single dose 0.045 mg/kg IV infused over 40 minutes
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — single dose 0.045 mg/kg IV infused over 40 minutes
  Arms: Midazolam
Drug: Ketamine — Single dose 0.5 mg/kg IV (in the vein) infused over 40 minutes
  Other Names: Racemic ketamine hydrochloride
  Arms: Ketamine

SUMMARY:
The objective of the proposed study is to test if a single IV dose of ketamine (0.5 mg/kg) decreases symptoms of PTSD.

DETAILED DESCRIPTION:
PTSD is a debilitating anxiety disorder characterized by intrusive re-experiences of the traumatic events, avoidance of situations and stimuli that could serve as reminders of these events, and feeling jumpy or easily startled. Patients with PTSD are often also depressed, and many have significant memory impairments. Existing drug treatments are unsuccessful in a majority of patients, especially in those with combat-related PTSD.

Our aim is to test the effectiveness of a potential new drug for PTSD, ketamine. For many years, intravenous ketamine has been extensively used for anesthesia. More recently, using doses lower than those used in anesthesia, a single ketamine infusion was shown to rapidly reduce depressed mood as well as anxiety in patients with severe depression. Some clinical evidence of potential efficacy in depressed patients with co-morbid PTSD also exists.

Adverse effects in these studies have been limited to feeling intoxicated and having increased blood pressure during the infusion.

In the present study, we expect a single ketamine infusion to reduce core PTSD symptoms. In addition, in those patients with PTSD who are depressed, we expect ketamine to reduce depressed mood.

Finally, ketamine is known to impair memory function temporarily. We will also test if the extent of ketamine-induced memory impairment during the infusion can predict how well people do after the infusion. Forty patients with PTSD (with and without combat-related trauma histories) will be tested, using a design that will compare the effectiveness of intravenous ketamine to that of midazolam, another anesthetic drug without any known long-term effects on anxiety, depressed mood, and memory function. If ketamine is found to have the expected effects, future studies may explore additional benefits of repeated infusions and / or alternatives to intravenous drug administration. Our study may contribute to improved function of patients with PTSD by providing a new means to rapidly treat their debilitating symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 21-55 years of age;
* Participants must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign a written informed consent document;
* Participants must fulfill DSM-IV criteria for current civilian or combat-related PTSD, based on clinical assessment by a study psychiatrist and on the CAPS (score must be at least 50 at screening and prior to each infusion - this is done to ensure at least moderate severity and to safeguard against high placebo response rates); additionally, clinicians will use clinical judgment to assess if patients are symptomatic enough to receive each infusion
* Women must be using a medically accepted reliable means of contraception (if using an oral contraceptive medication, they must also be using a barrier contraceptive) or not be of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year);
* Women of childbearing potential must have a negative pregnancy test at screening and pre-infusion;
* Participants must be able to identify a family member, physician, or friend (i.e. someone who knows them well) who will participate in a Treatment Contract (and e.g. contact the study physician on their behalf in case manic symptoms or suicidal thoughts develop).

Exclusion Criteria:

* Women who plan to become pregnant, are pregnant or are breast-feeding (because the medical risk of using ketamine during pregnancy and breast-feeding is unknown);
* Serious, unstable medical illnesses such as hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease (including gastro-esophageal reflux disease, obstructive sleep apnea, history of difficulty with airway management during previous anesthetics, ischemic heart disease and uncontrolled hypertension, and history of severe head injury);
* Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG;
* Patients with uncorrected hypothyroidism or hyperthyroidism;
* Hormonal treatment (e.g., estrogen) started in the 3 months prior to the first infusion day;
* Use of evidence-based individual psychotherapy (such as prolonged exposure) and other non-pharmacological treatments during the study;
* Histories of autism, mental retardation, pervasive developmental disorders, or Tourette's syndrome;
* History of one or more seizures without a clear and resolved etiology;
* History of (hypo)mania;
* Past or current presence of psychotic symptoms, or diagnosis of a lifetime psychotic disorder including schizophrenia or schizoaffective disorder;
* Drug or alcohol abuse or dependence within the preceding 3 months (given that this might otherwise contribute to their symptoms, however, a rather narrow time period was chosen such as to allow participation by individuals with a history of substance abuse or dependence problems that could be secondary to their PTSD, and to more closely approximate patients seen in real-world settings);
* Previous recreational use of ketamine or PCP;
* Current diagnosis of bulimia nervosa or anorexia nervosa;
* Diagnosis of schizotypal or antisocial personality disorder (since these are known to reduce the possibility of study completion; other Axis II diagnoses will be allowed);
* Patients judged clinically to be at serious and imminent suicidal or homicidal risk.
* A blood pressure of one reading over 160/90 or two separate readings over 140/90 at screen or baseline visits.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Charney, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Derived] Feder A, Parides MK, Murrough JW, Perez AM, Morgan JE, Saxena S, Kirkwood K, Aan Het Rot M, Lapidus KA, Wan LB, Iosifescu D, Charney DS. Efficacy of intravenous ketamine for treatment of chronic posttraumatic stress disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Jun;71(6):681-8. doi: 10.1001/jamapsychiatry.2014.62. PMID 24740528

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with chronic PTSD related to a range of trauma exposures were recruited via advertisements beginning Jan 2009, and were enrolled at the Icahn School of Medicine at Mount Sinai, New York, between May 2009 and December 2012.
Groups:
- Ketamine Then Midazolam: Ketamine: Single dose 0.5 mg/kg IV (in the vein) infused over 40 minutes on day 1,
  then 2 weeks later, Midazolam: single dose 0.045 mg/kg IV infused over 40 minutes
- Midazolam Then Ketamine: Midazolam: single dose 0.045 mg/kg IV infused over 40 minutes on day 1, then 2 weeks later, Ketamine: Single dose 0.5 mg/kg IV (in the vein) infused over 40 minutes
Period: First Infusion Day 1
Arm/Group | Ketamine Then Midazolam | Midazolam Then Ketamine
Started | 22 | 19
Completed | 22 | 19
Not Completed | 0 | 0
Period: no Infusion at Week 1
Arm/Group | Ketamine Then Midazolam | Midazolam Then Ketamine
Started | 22 | 19
Completed | 22 | 15
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — delayed-onset sedation | 0 | 1
Not completed — low baseline PTSD symptoms level | 0 | 1
Period: Second Infusion at 2 Weeks
Arm/Group | Ketamine Then Midazolam | Midazolam Then Ketamine
Started | 16 (N=6 completed the study at 2 wks due to CAPS scores < 50, precluding 2nd infusion.) | 15
Completed | 16 | 13
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — pt felt uncomfortable after infusion | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Midazolam the Ketamine: Midazolam: single dose 0.045 mg/kg IV infused over 40 minutes on Day 1, then 2 weeks later Ketamine: Single dose 0.5 mg/kg IV (in the vein) infused over 40 minutes
- Total: Total of all reporting groups
Arm/Group | Ketamine Then Midazolam | Midazolam the Ketamine | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (10.8) | 35.7 (10.0) | 36.05 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 9 | 13 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 12 | 23
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 11
Education [Number; unit: participants]
  less than high school | 1 | 0 | 1
  high school graduate | 3 | 3 | 6
  some college | 12 | 14 | 26
  more than 4 years of college | 5 | 2 | 7
  unknown | 1 | 0 | 1
Percentage Unemployed [Number; unit: percentage of participants] | 50 | 73.7 | 123.7
Primary Trauma [Number; unit: participants]
  Sexual assault or molestation | 9 | 0 | 9
  Physical assault or abuse | 4 | 7 | 11
  Accident or fire | 1 | 3 | 4
  Combat exposure | 2 | 0 | 2
  Witnessed violent assault or death | 4 | 5 | 9
  Witnessed 9/11 terrorist attacks | 2 | 0 | 2
  Unknown | 0 | 4 | 4
Duration of PTSD [Mean (Standard Deviation); unit: years] | 14.2 (12.3) | 11.9 (14.0) | 13.1 (13.1)
History of treatment with psychotropic medication [Number; unit: percentage of participants] | 50 | 42.1 | 92.1
Clinician-Administered PTSD Scale (CAPS) score (past month) [Mean (Standard Deviation); unit: units on a scale] — frequency score - scale 0 = none of the time to 4 = most or all of the time intensity score - scale 0 = none to 4 = extreme To meet criteria for a symptom, a patient must meet criteria in both frequency and intensity score for each item. Frequency and intensity and then combined to form a single severity score.
  30 questions scale, with total score ranging from 0 to 240.
  units on a scale | 82.5 (14.1) | 77.1 (11.8) | 80.0 (13.0)
Quick Inventory of Depressive Symptomatology, Self-Report (QIDS-SR) score [Mean (Standard Deviation); unit: units on a scale] — Each item is rated 0 (no depression) to 3 (severe depression). The total score ranges from 0-27.
  units on a scale | 12.4 (5.2) | 11.3 (5.6) | 11.9 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Impact of Event Scale - Revised (IES-R)
Description: A 22-item self-report questionnaire measuring PTSD symptoms. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score ranging from 0 (not at all) to 88 (extremely)
Time Frame: 7 days after first infusion
Population: Not all participants returned for the 1 week follow up visit. There were 19 participants from the Ketamine group and 15 participants from the Midazolam group who returned for their followup visit and completed the IES-R at the 1 week follow up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 19 | 15
units on a scale | 25.76 (19.4) | 36.32 (13.73)

2. Secondary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: Clinician-administered structured interview measuring PTSD symptoms. frequency score - scale 0 = none of the time to 4 = most or all of the time intensity score - scale 0 = none to 4 = extreme To meet criteria for a symptom, a patient must meet criteria in both frequency and intensity score for each item. Frequency and intensity and then combined to form a single severity score. 30 questions scale, with total score ranging from 0 to 240.
Time Frame: 7 days after first infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 19 | 15
units on a scale | 54 (23.63) | 65.69 (16.36)

3. Secondary Outcome: Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR)
Description: Self-report questionnaire measuring depressive symptoms. Each item is rated 0 (no depression) to 3 (severe depression). The total score ranges from 0-27.
Time Frame: 24 hours after first infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 22 | 19
units on a scale | 12.4 (5.2) | 11.3 (5.6)

4. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Clinician-administered questionnaire measuring depressive symptoms. The MADRS-S has 10-items which are based on mood symptoms over the past 7 days. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression). Mean difference between baseline and 2 weeks.
Time Frame: 24 hours after first infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 22 | 19
units on a scale | 12.6 (7.9) | 10.1 (9.7)

5. Secondary Outcome: Hopkins Verbal Learning Test (HVLT)
Description: Repeatable test of memory acquisition and delayed recall of words. It is a three-trial list learning and free recall task comprising 12 words, 4 words from each of three semantic categories. Total Recall score range is 0 to 36.
Time Frame: 20 to 40 minutes after infusion
Population: data not collected
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours post infusion
Groups:
- Ketamine: Ketamine: Single dose 0.5 mg/kg IV (in the vein) infused over 40 minutes,
Arm/Group | Ketamine | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/31
Serious Adverse Events (participants affected / at risk) | 33/38 | 31/31
Other Adverse Events (participants affected / at risk) | 0/38 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=38) | Midazolam (N=31)
Diarrhea (Gastrointestinal disorders) | 3 | 2
Dry Mouth (Gastrointestinal disorders) | 10 | 4
Nausea/Vomiting (Gastrointestinal disorders) | 10 | 0
Palpitation (Cardiac disorders) | 3 | 0
Dizziness on standing (Cardiac disorders) | 6 | 5
Chest Pain (Cardiac disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Increased perspiration (Skin and subcutaneous tissue disorders) | 3 | 1
Itching (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Headace (Nervous system disorders) | 8 | 4
Tremors (Nervous system disorders) | 0 | 1
Poor coordination (Nervous system disorders) | 7 | 1
Dizziness (Nervous system disorders) | 14 | 9
Blurred vision (Eye disorders) | 15 | 6
Ringing in ears (Ear and labyrinth disorders) | 5 | 1
Difficulty urinating (Renal and urinary disorders) | 0 | 3
Painful urination (Renal and urinary disorders) | 2 | 1
Frequent urination (Renal and urinary disorders) | 2 | 4
Difficulty sleeping (General disorders) | 3 | 3
Sleeping too much (General disorders) | 2 | 1
Anxiety (General disorders) | 5 | 1
Poor concentration (General disorders) | 4 | 6
General malaise (General disorders) | 3 | 1
Restlessness (General disorders) | 13 | 4
Fatigue (General disorders) | 10 | 6
Decreased energy (General disorders) | 6 | 3

LIMITATIONS AND CAVEATS:
Several patients did not receive a second infusion per protocol because of sustained reduction in PTSD symptom levels . The study also does not address the safety or efficacy of ketamine in combination with other psychotropic medications in PTSD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes